CLINICAL TRIAL: NCT02927379
Title: Effects of Local Wound Infiltration With Ketamine Versus Dexmedetomidine Added to Bupivacaine on Surgical Stress Response and Postoperative Pain in Major Abdominal Cancer Surgery
Brief Title: Effect of Wound Infiltration by Ketamine Versus Dexmedetomidine Added to Bupivacaine on Surgical Stress
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fatma Adel El sherif, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 248
Record Dates: First submitted 2016-10-05; First posted 2016-10-07 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2017-06

CONDITIONS: Abdominal Cancer
MeSH Terms: interventions — Dexmedetomidine; Injections, Subcutaneous; Ketamine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ketamine group (Active Comparator): intervention: local wound infiltration 30 patients receive local anesthetic wound infiltration with with 20 ml of bupivacaine 0.5 % diluted in 20 ml saline +1 mg /kg ketamine (total volume 40 ml) in two divided doses i.e. 20 ml is administered on each side of incision.
  Interventions: Drug: Ketamine
- dexmedetomidine group (Active Comparator): intervention: local wound infiltration 30 patients receive local anesthetic wound infiltration with with 20 ml of bupivacaine 0.5 % diluted in 20 ml saline + 1µg/kg dexmedetomidine (total volume 40 ml) in two divided doses i.e. 20 ml is administered on each side of incision.
  Interventions: Drug: Dexmedetomidine
- bupivacaine group (Placebo Comparator): intervention: local wound infiltration 30 patients receive local anesthetic wound infiltration with with 20 ml of bupivacaine 0.5 % diluted in 20 ml saline (total volume 40 ml) in two divided doses i.e. 20 ml is administered on each side of incision( control group).
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Dexmedetomidine — local anesthetic wound infiltration with with 20 ml of bupivacaine 0.5 % diluted in 20 ml saline plus dexmetedomidine in two divided doses i.e. 20 ml is administered on each side of incision
  Other Names: subcutaneous
  Arms: dexmedetomidine group
Drug: Ketamine — local anesthetic wound infiltration with with 20 ml of bupivacaine 0.5 % diluted in 20 ml saline plus ketamine in two divided doses i.e. 20 ml is administered on each side of incision
  Other Names: subcutaneous
  Arms: ketamine group
Drug: Bupivacaine — local anesthetic wound infiltration with with 20 ml of bupivacaine 0.5 % diluted in 20 ml saline only in two divided doses i.e. 20 ml is administered on each side of incision
  Other Names: subcutaneous
  Arms: bupivacaine group

SUMMARY:
This study aims to compare the effects of local wound infiltration with ketamine versus dexmedetomidine when added to bupivacaine on stress response and postoperative pain in lower abdominal cancer surgery.

DETAILED DESCRIPTION:
Patients will be randomly assigned using an online research randomizer into three groups, 30 patients in each group:

Group C:

30 patients receive local anesthetic wound infiltration with with 20 ml of bupivacaine 0.5 % diluted in 20 ml saline (total volume 40 ml) in two divided doses i.e. 20 ml is administered on each side of incision( control group).

Group K:

30 patients receive local anesthetic wound infiltration with with 20 ml of bupivacaine 0.5 % diluted in 20 ml saline +1 mg /kg ketamine (total volume 40 ml) in two divided doses i.e. 20 ml is administered on each side of incision.

Group D:

30 patients receive local anesthetic wound infiltration with with 20 ml of bupivacaine 0.5 % diluted in 20 ml saline + 1µg/kg dexmedetomidine (total volume 40 ml) in two divided doses i.e. 20 ml is administered on each side of incision.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) class I-II Body weight of 50 - 90 kg

Exclusion Criteria:

* History of bleeding diathesis
* Relevant drug allergy, opioid dependence
* Morbid obesity, sepsis

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2016-06; Primary Completion 2016-12 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Total morphine consumption | 24 hours

SECONDARY OUTCOMES:
Plasma concentrations of prolactin, cortisol and glucose level | 24 hours
the severity of pain was assessed using VAS score | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: fatma A EL sherif, Principal Investigator — South Egypt Cancer Instuite, Assuit, Assuit university
Locations (1):
- South Egypt Cancer Instuite, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mohamed SA, Sayed DM, El Sherif FA, Abd El-Rahman AM. Effect of local wound infiltration with ketamine versus dexmedetomidine on postoperative pain and stress after abdominal hysterectomy, a randomized trial. Eur J Pain. 2018 May;22(5):951-960. doi: 10.1002/ejp.1181. Epub 2018 Feb 1. PMID 29388288